CLINICAL TRIAL: NCT04030286
Title: Analysis of Serum and Salivary Malondialdehyde and Lipid Profile Levels in Patients With Periodontal and Cardiovascular Diseases
Brief Title: Evaluation of Malondialdehyde in Periodontal and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Junior Assistant Professor, University of Messina
Other Study IDs: 16-12
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Healthy patients
  Interventions: Other: Observation
- Periodontitis: Patients with periodontal disease
  Interventions: Other: Observation
- Cardiovascular: Patients with cardiovascular disease
  Interventions: Other: Observation
- Periodontitis+Cardiovascular: Patients with both periodontal and cardiovascular disease
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Evaluation of Malondialdehyde level and correlation of Malondialdehyde level with periodontal and cardiovascular disease

SUMMARY:
Malondialdehyde (MDA) plays a key role in endothelial function and may be a link for the known interaction of periodontitis and coronary heart disease (CHD). The investigators compared the impact of gingival health, periodontitis (CP), CHD or of both diseases (CP+CHD) on saliva and serum MDA levels.

DETAILED DESCRIPTION:
The aim of this study was to evaluate a possible association between both saliva and serum MDA levels in patients with CP and with CHD and if the serum MDA levels are mediated by serum CRP

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least twenty teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 32 healthy subjects, 34 patients with CP, 33 patients with CHD and 34 patients with CP and CHD. Lipid profile and levels of MDA and C-reactive protein (CRP) were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde levels | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol